CLINICAL TRIAL: NCT04856332
Title: VIK-e2 - Observational, Multicenter Prospective Study Evaluating Parent-child Relationship with the Setting Up of a Mobile Telepresence Robot for Patients with Children Aged 15 Years or Less and Hospitalised in Long-term Protective Isolation
Brief Title: Study Evaluating the Parent-child Relationship During the Hospitalisation of a Parent in Long-term Protective Isolation
Acronym: VIK-e2
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET19-193 - VIK-e2
Record Dates: First submitted 2021-04-08; First posted 2021-04-23 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: Cancer; Long-term protective isolation; Patient-child relationship
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Telepresence robot installed at child's home during parent's hospitalisation — Telepresence robot installed at child's home during parent's hospitalisation in long term protective isolation for maintaining parent-child ink (only children aged 15 years or less are concerned)

SUMMARY:
The intensive treatments of certain cancers and haemopathies require the implementation of a protective isolation from external micro-organisms for a period of several weeks. This isolation implies a limitation of visitors and sometimes prohibits access to young children. This raises questions concerning the maintenance of family links, and in particular the parent-child relationship as well as the psychological and emotional isolation of hospitalised patients and the resulting psychological effects.

DETAILED DESCRIPTION:
Telepresence robots are increasingly used as a means of remote communications, especially for teleconsultations and/or access to various public services (cultural events, education, etc.). In the context of long-term hospitalisation, they can be used for various purposes, such as access to cultural events, university activities, contact with patient's home and maintenance of family links. Some studies have analyzed the use of these robots and their effects in academic settings or the suitability of their use with elderly populations for continuing care.

To our knowledge, no study has evaluated the interest for the parent-child relationship of the use of a telepresence robot during the hospitalisation in protective isolation for a long period of a patient with young child(ren).

We propose to conduct this observational, multi-center prospective study aiming at evaluating the parent-child relationship following the setting up of a mobile telepresence robot for patients with children aged 15 years or less and hospitalised in long-term protective isolation.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18
* Patient with at least one child aged 15 or under
* Pathology requiring a prolonged hospitalization in protective isolation
* Consent dated and signed

Exclusion Criteria:

* Impaired cognitive functions
* Performance Status -Eastern Cooperative Oncology Group (PS-ECOG) = 4
* Difficulties in speaking and understanding French
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Observational prospective study, multicenter of parent-child relationship assessment following the setting up of a mobile telepresence robot for patients with children aged 15 years or less and hospitalised in long-term protective isolation. This study is based on semi-directed interviews and observations made during patient's hospitalisation and when patient returns at home.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the use of a telepresence robot on the parent-child relationship in maintaining parenthood during parent's hospitalisation in long-term protective isolation | Through study completion, an average of 3 months
  Observation of communications between the hospitalised patient and his/her chid(children) by a specialist in human and social sciences
Evaluation of the use of a telepresence robot on the parent-child relationship in maintaining parenthood during parent's hospitalisation in long-term protective isolation | Through study completion, an average of 3 months
  Interview with the hospitalised patient (parent) by a specialist in human and social sciences

SECONDARY OUTCOMES:
Evaluation of the experience linked to the robot availability on the concerned persons (patient, children, person on charge of children) | Through study completion, an average of 3 months
  Interview with the hospitalised patient (parent) and the person in charge of children by a specialist in human and social sciences
Evaluation of patient's satisfaction | Through study completion, an average of 3 months
  Interview with the hospitalised patient (parent) and the person in charge of children by a specialist in human and social sciences
Evaluation of the impact of robot use on patient's coping strategies (adaptation and adjustment to illness and hospitalisation) | Through study completion, an average of 3 months
  Interview with the hospitalised patient and the person in charge of children by a specialist in human and social sciences
Evaluation of patient's experience of hospitalisation | Through study completion, an average of 3 months
  Interview with the hospitalised patient and the person in charge of children by a specialist in human and social sciences
Evaluation of the impact of the robot's presence at home on the children and the person in charge of the children during patient's hospitalisation | Through study completion, an average of 3 months
  Interview with the hospitalised patient and the person in charge of children by a specialist in human and social sciences

CONTACTS AND LOCATIONS:
Overall Officials: GUILLERMIN Yann, MD, Principal Investigator — Centre Leon Berard
Locations (3):
- France (3):
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Lyon Sud, Lyon
  - Institut Paoli Calmettes, Marseille